**Document Type:** Informed Consent Form

Official Title: Effect of Dietary Advice Source on Perceptions of Information Accuracy and Intended

Compliance

NCT Number: NCT04858971

**IRB Approval Date:** 07/12/2021

# GRAND FORKS HUMAN NUTRITION RESEARCH CENTER CONSENT TO PARTICIPATE IN RESEARCH

Project Title: Survey of Diet and Health Beliefs

Principal Investigators: Alese M. Nelson, Ph.D., James Roemmich, Ph.D.

Email Addresses: alese.nelson@usda.gov

#### What should I know about this research?

• Taking part in this research is voluntary. Whether you take part is up to you.

- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you.
- If you don't understand, ask questions. You may contact the researchers above with questions before you consent to the study.
- Ask all the questions you want before you decide.

# How long will I be in this research?

We expect that your taking part in this research will last about one (1) hour. You will be asked to answer around 200 questions. The exact number of questions you answer will depend on your responses, as some questions may have follow-up questions based on how you respond.

#### Why is this research being done?

The purpose of this research is to better understand people's health and diet knowledge, beliefs, attitudes, and practices. We will use this information to implement better strategies to help Americans maintain more nutritious diets.

#### What happens to me if I agree to take part in this research?

If you decide to take part in this research study, you will fill out a series of questionnaires. These questions will be about you: your demographic information, your beliefs, your attitudes, your knowledge, and your practices.

Some of these questions will be personal. If you feel uncomfortable answering any of these questions, you are free to skip them or select the box that says, "prefer not to answer," if available. You will also see a health information flyer and will be asked to provide feedback regarding your opinions of the flyer.

#### Could being in this research hurt me?

The risks or discomforts that you may experience from taking part in this research include psychological and/or emotional discomfort because of being asked personal questions.

Additionally, because this research is conducted online, there is always the possibility of a security breach. Given that surveys can be completed from any computer (e.g., personal, work, school), we are unable to guarantee the security of the computer on which you choose to enter your responses. As a participant in our study, we want you to be aware that certain 'key logging' software programs exist that can be used to track or capture data that you enter and/or websites that you visit. To minimize your risk, we recommend that you complete this survey on a private device connected to a private, secure network. Although every reasonable effort has been taken, confidentiality during actual Internet communication procedures cannot be guaranteed.

#### Will being in this research benefit me?

It is not expected that you will personally benefit from this research, though you may also gain personal insights because of answering these questions. Possible benefits to others include increased knowledge and understanding of how to improve health.

#### How many people will participate in this research?

We expect 1000 people will complete this study conducted by the Grand Forks Human Nutrition Research Center.

#### Will it cost me money to take part in this research?

You will not have any costs for being in this research study.

# Will I be paid for taking part in this research?

You will be paid for being in this research study. You will receive a payment of \$45 through your Amazon Mechanical Turk account within 5 days of your completion of the study (i.e., submission of the survey).

To protect the integrity of our research, <u>each person is limited to one completion</u> of this survey. If you attempt this survey more than once, you <u>will not</u> receive payment for additional completions. Researchers will review responses to ensure they come from unique individuals. Furthermore, it is important that participants read the survey questions and respond truthfully. Researchers will review responses for suspicious activity. If a survey response is flagged for bad responses (for example, clicking through rather than providing genuine responses), you <u>will not</u> receive payment.

Please note: While you are welcome to skip questions that make you uncomfortable, to receive payment for this survey, we need participants to complete at least 90% of the survey. We will review surveys prior to approving payment to ensure the survey was at least 90% completed. If you have skipped less than 20 questions/responses, you can expect to receive payment within 5 days of completing the survey. If you skipped more than 20 questions/responses, you would <u>not</u> receive payment. If you have concerns regarding the number of questions you skipped, please contact Alese Nelson (alese.nelson@usda.gov).

#### Who is funding this research?

This research is being funded by the Grand Forks Human Nutrition Research Center (GFHNRC), a branch of the United States Department of Agriculture, Agricultural Research Service (USDA ARS). This means that the GFHNRC is receiving payments from the USDA to support the activities that are required to conduct this study. No one on the research team will receive a direct payment or an increase in salary from the USDA for conducting this study.

# What happens to information collected for this research?

Your private information may be shared with individuals and organizations that conduct or watch over this research, including:

- The researchers
- People who work with the researchers (support staff)
- The United States Department of Agriculture Agricultural Research Service
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep any identifying information confidential. We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy.

Data collected in this research might be de-identified and used for future research or distributed to another investigator for future research without your consent.

## What if I agree to be in the research and then change my mind?

If you decide to leave the study early, we ask that you send an email to <u>alese.nelson@usda.gov</u> to notify us of your withdrawal. You may stop the survey at any time.

#### Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the email address listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at 701.777.4279 or <a href="https://www.undies.com/undie

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.
- You may also visit the UND IRB website for more information about being a research subject: <a href="http://und.edu/research/resources/human-subjects/research-participants.html">http://und.edu/research/resources/human-subjects/research-participants.html</a>

Checking this box documents your consent to take part in this study.

By checking this box, I certify that:

- I am 18 years old or older.
- I am a U.S. citizen.
- · I have read and agree to the terms above.
- · I freely consent to participate in this study.
- ☐ I am at least 18 years old, a U.S. citizen, I have read and agree to the terms above, and I freely consent to participate in this study.